CLINICAL TRIAL: NCT00220116
Title: A Phase II Trial Assessing the Efficacy and Toxicity of Capecitabine and Oxaliplatin in the Treatment of Colorectal Cancer.
Brief Title: Phase II Trial Assessing Efficacy and Toxicity of Capecitabine and Oxaliplatin in the Treatment of Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Jane Lawrence, Royal Marsden NHS Foundation Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2147
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2010-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Capecitabine, Oxaliplatin

SUMMARY:
To assess the efficacy and safety of the combination of capecitabine and oxaliplatin in the 1st, 2nd or subsequent line treatment of metastatic colorectal cancer, and also in the neo-adjuvant and adjuvant setting of resectable metastases.

Primary Endpoint: Objective response rates

Secondary Endpoints: Treatment related toxicity Progression free survival (If not resected) Disease free Survival (From metastastectomy, if resected) Overall Survival 60 Day all cause mortality Number undergoing liver resections/curative resection (Ro) rate

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Histologically proven colorectal adenocarcinoma, requiring therapy as defined by one of the four treatment subgroups
* No previous malignant disease other than non-melanotic skin cancer or carcinoma-in-situ of the uterine cervix.
* Unidimensional measurable disease as assessed by CT. (Unless adjuvant therapy only)
* Adequate bone marrow function; Hb >10g/dl, platelets >100 x109/l, WBC >3x109/l, Neut >1.5x109/l.
* Adequate liver function: Serum Bilirubin <1.5 x upper limit of institutional normal
* Adequate renal function, calculated Creatinine Clearance >50mls/min
* No concurrent uncontrolled medical conditions
* WHO performance status 0,1 or 2
* Adequate contraceptive precautions, if appropriate
* Informed written consent
* Negative pregnancy test in women of child bearing age
* Life expectancy > 3 months

Exclusion Criteria:

* Medical or psychiatric condition that comprise the patient's ability to take informed consent.
* Clinically significant (i.e. active) cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmia even if controlled with medication) or myocardial infarction within the last 12 months.
* Patients with any significant symptoms or history of peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2002-08

PRIMARY OUTCOMES:
Objective response rates

SECONDARY OUTCOMES:
Treatment related toxicity
Progression free survival (If not resected)
Disease free Survival (From metastastectomy, if resected)
Overall Survival
60 Day all cause mortality
Number undergoing liver resections/curative resection (Ro) rate

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital, Sutton, Surrey, United Kingdom